CLINICAL TRIAL: NCT05592119
Title: Effect of Stimulant Medication on Loss of Control Eating in Youth With Attention Deficit/Hyperactivity Disorder: a Prospective, Observational Case Series
Brief Title: Effect of Stimulant Medication on Loss of Control Eating in Youth With Attention Deficit/Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Aaron Keshen, Dr. Aaron Keshen, MD, FRCPC, Nova Scotia Health Authority
Other Study IDs: 1028376
Record Dates: First submitted 2022-10-14; First posted 2022-10-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Loss of Control Eating; Attention Deficit/Hyperactivity Disorder
Keywords: Stimulants; Eating disorders; Children; Binge eating
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Feeding and Eating Disorders; Bulimia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Loss of control eating (LOC-E) in youth predicts the later development of full syndrome eating disorders, such as binge-eating disorder (BED), and therefore, could be a relevant target for prevention interventions. Children with attention deficit/hyperactivity disorder (ADHD) are at higher risk of experiencing LOC-E than healthy controls, and there is evidence that related neurocognitive predisposing factors, such as impulsivity and dysfunctional reward processing, are associated with the pathogenesis of LOC-E. Therefore, it is pertinent to examine whether modifying these neurocognitive symptoms influences LOC-E and the subsequent development of eating disorders. Stimulants are an efficacious treatment for impulsivity in youth with ADHD and have been shown to improve symptoms of binge eating in adults; however, studies have not prospectively explored the effect of stimulants on LOC-E in youth. To explore this gap, the investigators aim to collect prospective observational data in a clinical setting to measure change in LOC-E episodes and secondary outcomes in youth aged 8 to 13 years old with ADHD and LOC-E who are treated with stimulants. The investigators will collect outcome measures prior to stimulant initiation (baseline) and 3 months after stimulant initiation.

DETAILED DESCRIPTION:
This study will use a prospective, observational case series design. Participants will be a prospective cohort sample of males and females aged 8 to 13 years old, and their parents/guardians, who have been referred to either: a) the Atlantic ADHD Centre in Dartmouth, Nova Scotia; b) the Mill Cove Medical Pediatric Clinic in Bedford, Nova Scotia; c) the general pediatrics outpatient clinic at IWK in Halifax, Nova Scotia; or d) the Beyond ADHD virtual clinic based out of New Brunswick. The research team will be based out of the Nova Scotia Health Authority Eating Disorder Clinic (Abbie J Lane Building; QEII Health Sciences Centre) in Halifax, Nova Scotia.

Due to the duration and limited success of recruitment, our team has decided to decrease the sample size. As of June 2024, our study will decrease from an estimated sample size of 40 parent-child pairs (80 total participants) to 10 (20 total). This will allow us to complete the study within the expected timeline and design a study that addresses the slower than expected recruitment (e.g., expand future recruitment sites).

Clinicians in the Atlantic ADHD Centre routinely pre-screen for LOC-E, using the Child Brief Binge-Eating Questionnaire (CBBEQ; Franklin et al., 2019), as part of their standard clinical assessment (see Appendix for schedule of assessments). This assessment also includes a psychiatric history by an ADHD expert and cognitive data using a validated Continuous Performance Test (CPT). Patients who are diagnosed with ADHD and pre-screen positive for LOC-E (score of 8 or above on CBBEQ), and who receive a recommendation to start a stimulant medication and intend to initiate the stimulant, will be invited to a consent and screening visit. Prescreening data collection is standard practice at the centre (i.e., relevant personal health information and scale-based outcomes) and will not be recorded for the study, as consent will not have been obtained. However, clinic staff will record the following non-personal health information that can be used in a participant flow diagram for study purposes: a) number of positive and negative pre-screens, and b) number of patients who are interested or not interested in being contacted by a research team member to learn more about the study.

At the clinics, parents/guardians and children who are interested in participating will be provided with an information sheet about the study. The parent/guardian will be asked to provide written consent to be contacted via their email or telephone by the research team. Parents/guardians who consent to being contacted will be sent a link to the electronic consent form (on REDCap). Once they have reviewed and signed the consent form, they will be asked to answer screening questions about their child (see Inclusion/Exclusion Criteria below). The parent/guardian of eligible potential child participants will be contacted about booking a Screening/Baseline interview, which will be held via Zoom for Healthcare or in-person at the Nova Scotia Health Authority Eating Disorder Clinic.

After a child is diagnosed with ADHD, clinicians at the Mill Cove Medical Pediatric Clinic, the general pediatrics outpatient clinic at IWK, and Beyond ADHD generally prescribe stimulant medications themselves. At the Atlantic ADHD Centre, children are referred back to their general practitioner to initiate a stimulant medication. If a child's scheduled appointment with their general practitioner to initiate a stimulant (which will occur naturalistically outside of the study context) is >2 weeks away, they will complete an initial Screening interview with a research assistant, and if they are found eligible a separate Baseline interview will be booked within 1-2 weeks of their appointment with the general practitioner. Child participants who are scheduled to see their general practitioner within the next 1-2 weeks will complete the Screening and Baseline measures with a research assistant within the same interview, provided they are found eligible after the screening portion of the interview.

At the start of the Screening interview, a research assistant will review the informed consent form with parent/guardian. Verbal consent to participate will be obtained from the parent/guardian. Then, the research assistant will conduct the assent discussion with the child, by following the Assent Script, and will complete the Assent Form. Verbal assent to participate will be obtained from the child.

This study will obtain baseline and outcome measurements through a series of assessments at 2 time-points: prior to initiating a stimulant (i.e., Baseline) and 3-months post initiation (i.e., follow-up). These assessments will be administered by a trained research assistant.

Means and standard deviations were calculated at both baseline and follow-up for primary and secondary objectives. In addition, mean reductions were calculated by subtracting the baseline and follow-up mean scores. Descriptive statistics (e.g., means and standard deviations) will be used to report demographic information, medication doses, adverse events, and frequency of medication discontinuation. If available, reasons for medication discontinuation and loss to follow-up will be documented. Given the case series design, there will be no a priori power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Youth 8 to 13 years of age
* Able to provide informed consent
* Meet DSM-V diagnostic criteria for ADHD
* Experienced at least 3 episodes of LOC-E during the past 3 months, accompanied by some degree of distress and 2 of the 5 behavioural symptoms associated with LOC-E

Exclusion Criteria:

* Currently receiving treatment for overweight
* Taking medication with effects on eating behaviour
* Insufficient English language skills

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female youth aged 8 to 13 years old who are diagnosed with ADHD and LOC-E at the Atlantic ADHD Centre in Dartmouth, Nova Scotia.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Change in LOC-E episode frequency | Screening, Baseline, 3 Months
  This will be measured using the Child Version of the Eating Disorder Examination (ChEDE C.1; Bryant-Waugh et al., 1996; Bryant-Waugh, 2020). The EDE 17.0D (Fairburn et al., 2014), which measures eating disorder symptom severity, has been modified for use with children ages 8 and above (Bryant-Waugh et al., 1996; Bryant-Waugh, 2020). The ChEDE has been shown to have high inter-rater reliability and internal consistency (Hilbert et al., 2013; Watkins et al., 2005). For the purposes of this study, only diagnostic item 11 (identifying bulimic episodes and other episodes of overeating) of the ChEDE will be used, which included questions regarding feelings of loss of control eating, features associated with binge eating, and distress about binge eating. The measure will be used for diagnostic assessment of LOC-E for study inclusion purposes, and at Baseline and 3-Month Follow-Up to establish LOC-E episode frequency.

SECONDARY OUTCOMES:
Change in eating behaviour | Baseline, 3 Months
  This will be measured at Baseline and 3-Month Follow-Up using the Child Eating Behaviour Questionnaire (CEBQ; Wardle et al., 2001). The CEBQ, to be completed by the parent/guardian, is a valid and reliable 35-item measured used to evaluate cognitions, emotions, and behaviors associated with disordered eating, rated on a 5-point Likert scale with scores ranging from 1 (never) to 5 (always). Higher scores indicate a greater global level of disordered eating (Wardle et al., 2001; Carnell & Wardle, 2007).
Change in disordered eating | Baseline, 3 Months
  This will be measured at Baseline and 3-Month Follow-Up using the Eating Disorder Examination Questionnaire adapted for children (ChEDE-Q8; Kliem et al., 2017).The ChEDE-Q8 is valid self-report version of the ChEDE, evaluating areas of eating disorder psychopathology, with scores on the 8-item measure ranging from 0 (absent) to 6 (extreme everyday presence) with high internal consistency (Kliem et al., 2017). Higher scores indicate higher levels of eating disorder psychopathology.
Change in ADHD symptom severity | Baseline, 3 Months
  This will be measured using the Vanderblit ADHD Diagnostic Parent Rating Scale (VADPRS; Wolraich et al., 2003), a 56-item measure used to evaluate ADHD behaviors, along with academic and social performance in children to be completed the parent/guardian. The ADHD symptoms has scores ranging from 0 (never) to 3 (very often) on a 4-point Likert scale, with higher scores indicating greater levels of ADHD behaviours. The performance component has scores ranging from 1 (excellent) to 5 (problematic) on a 5-point scale, with higher scores indicating greater impairment in academic and/or social performance. This will be administered at Baseline and with an adapted/shortened version at a 3-Month Follow-Up. The VADPRS has demonstrated good construct, discriminant, and content validity, as well as internal consistency (Wolraich et al., 2003; Collett et al., 2003; Wolraich et al., 2013; Bard et al., 2013).
Change in Impulsivity and reward sensitivity | Baseline, 3 Months
  This will be measured by the Parent-Report Behavioral Inhibition System/Behavioral Activation System Scales (BIS/BAS; Vervoort et al., 2015) at Baseline and 3-Month Follow-Up. This 20-item parent-report measure, which was adapted from the original self-report BIS/BAS scales (Carver & White, 1994), examines two motivational systems through responses to reward and punishment. Impulsivity has been found to be positively correlated with BAS-drive and BAS-fun seeking, and negatively correlated with BIS (Franken et al., 2005); therefore, the BIS/BAS can be used as a proxy for impulsivity in youth. Scores range from 1 (not true at all) to 4 (all true) on a 4-point Likert scale. The total separate scores of the four subscales will be used, with higher scores indicating greater levels of sensitivity in the associated motivational system. The parent-report BIS-BAS is a reliable and valid tool for examining punishment and reward sensitivity in children (Vervoort et al., 2015).
Change in anxiety/mood severity | Baseline, 3 Months
  This will be measured using the Revised Child Anxiety and Depression Scale - Short Version (RCADS-25; Ebesutani et al., 2012) at Baseline and 3-Month Follow-Up. This 25-item self-report measure, adapted from the original 47-item RCADS (Chorpita et al., 2000; Chorpita et al., 2005), is used to assess depression and anxiety symptoms in children. The RCADS-25 contains 10 questions based on major depressive disorder, and 15 questions based on five DSM-IV anxiety domains: separation anxiety disorder, generalized anxiety disorder, panic disorder, social phobia, and obsessive-compulsive disorder. RCADS-25 scores range from 0 (never) to 3 (always) on a 4-point Likert scale. Global anxiety and depression scores will be used separately, with higher scores on each scale indicating greater levels of anxiety and depression. The RCADS-25 is a reliable clinical tool and has been shown to have discriminant, convergent, and divergent validity (Ebesutani et al., 2017).
Parental/Guardian LOC-E | Baseline
  This will be measured using the LOCES (Latner et al., 2014), which is to be completed by parents/guardians at Baseline in relation to their own eating psychopathology. This 24-item self-report measure used to examine three aspects of LOC-E: behavioural, cognitive/dissociative, and positive/euphoric. The LOCES consists of three subscales based on the three aspects of LOC-E, with scores ranging from 1 (never) to 5 (always) on a 5-point Likert scale. The global mean score calculated from the average of each subscale will be used, with higher scores indicating greater levels of LOC-E. The LOCES has been shown to have high internal consistency, convergent and discriminant validity, and test-retest reliability (Latner et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Keshen, MD, FRCPC, Principal Investigator — Department of Psychiatry, Dalhousie University, Halifax, Nova Scotia
Locations (1):
- Abbie J Lane Memorial Building - QEII, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Keshen AR, Hilbert A, Taylor V, Harris AL, Trappenberg N, Sadek J, Frank GKW, Murray SB. Effect of stimulant medication on loss of control eating in youth with attention deficit/hyperactivity disorder: a prospective, observational case series study protocol. J Eat Disord. 2022 Nov 1;10(1):152. doi: 10.1186/s40337-022-00674-y. PMID 36320022